CLINICAL TRIAL: NCT03802955
Title: A Phase Ⅰ Study of ADG106 Administered in Patients With Advanced or Metastatic Solid Tumors and/or Non-Hodgkin Lymphoma
Brief Title: Study of ADG106 With Advanced or Metastatic Solid Tumors and/or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adagene (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: Adagene Inc (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG106-1002
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumor; Non-Hodgkin Lymphoma
Keywords: Solid Tumor; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADG106 Dose escalation (Experimental)
  Interventions: Drug: ADG106

INTERVENTIONS:
Drug: ADG106 — IV infusion over 60 minutes on Day 1 of each cycle, at 7 doses depending on cohort at enrollment.

SUMMARY:
This is a Phase 1, open-label, dose-escalation, single-center study of ADG106 in subjects with advanced or metastatic solid tumors and/or relapsed/ refractory non-Hodgkin lymphoma. ADG106 is a fully human ligand-blocking, agonistic anti-CD137 IgG4 mAb. It binds to the activated human T cells via a T cell receptor CD137. ADG106 administered intravenously (IV) over a period of 60-90 minutes.

Primary objective:

To assess safety and tolerability at increasing dose levels of single agent ADG106 in subjects with advanced or metastatic solid tumors and/or non Hodgkin lymphoma.

To determine the recommended dosage and dosage regimen for further study. Secondary Objectives To characterize the pharmacokinetic (PK) profiles of ADG106. To evaluate the immunogenicity of ADG106. To evaluate the potential anti-tumor effect of ADG106. To investigate serum biomarkers related to immune regulation and cytokine releasing.

Exploratory Objective:

To identify the potential biomarkers of ADG106.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years to 75 years of age at the time of consent.
2. Provide written informed consent.
3. Subjects with advanced and/or metastatic histologically or cytologically confirmed solid tumor and/or non-Hodgkin lymphoma who are refractory or relapsed from standard therapy and who have exhausted all available therapies.
4. At least one measurable lesion per RECIST 1.1 for solid tumors and per Lugano Classification for non-Hodgkin lymphoma
5. ECOG performance: 0-1
6. Adequate organ and bone marrow function
7. After receiving the last treatment (chemotherapy, radiotherapy, biotherapy or other research drugs), the patient had a washout period of at least 4 weeks or more than 5 half-lives, and had recovered from any toxic reaction of the previous treatment to less than 1 degree.
8. No other concomitant antineoplastic therapy (including cell therapy)
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within the 7 days prior to study drug administration.
10. Coagulation function is basically normal, INR≤1.5
11. Cooperative in observation of adverse events and efficacy

Exclusion Criteria:

1. Subjects with positive HCV antibody，or active hepatitis B (HBV DNA ≥ 10000 copies/mL or 2000 IU/mL), or positive hepatitis virus and taking antiviral drugs
2. Subjects with meningeal metastasis, or subjects with brain metastasis lesions ≥ 1 cm and untreated, or subjects with brain metastasis requiring mannitol or other dehydration therapy
3. Infection of human immunodeficiency virus (HIV), or suffering from other acquired, congenital immunodeficiency disorders, or organ transplantation history
4. Any active autoimmune disease or evidence-based autoimmune disease, or systemic syndrome requiring systemic steroids or immunosuppressive drugs (Except for inactive vitiligo, psoriasis, asthma/specific reactivity in children after treatment within two years, or thyroid diseases controlled by alternative therapy/non-immunosuppressive therapy）
5. The residual toxicity of the patient's previous treatment was more than grade 1
6. Fever body temperature above 38℃ or there are clinically obvious active infections that can affect clinical trials
7. Overdose of glucocorticoid (>10mg/d prednisone or equivalent dose) or other immunosuppressive agents was used within one month
8. According to the investigator, any uncontrollable serious clinical problems include but are not limited to, evidence of severe or uncontrollable systemic diseases (such as unstable or uncompensated respiratory, cardiac, liver or kidney diseases); and any unstable systemic diseases (including active infections, refractory high or drug failure Controlled hypertension (>150/100 mmHg), unstable angina pectoris, congestive heart failure, liver and kidney or metabolic diseases）
9. A clear history of neurological or psychiatric disorders, including epilepsy or dementia
10. Non-research-related surgical procedures performed prior to the use of research drugs in patients within 28 days
11. Investigator do not consider he/she appropriate to participate in this study
12. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
DLTs in the first 2 cycles of single drug administration | 2 Cycles (42 days)

SECONDARY OUTCOMES:
Number of clinical and laboratory adverse events (AEs) . | First dose to 30 days post last dose
Objective response rate (ORR) as assessed by RECIST version 1.1 and immune-related RECIST (irRECIST) for solid tumor and the Lugano Classification for non-Hodgkin Lymphoma | 2 Cycles (42 days)
Duration of response (DOR) as assessed by RECIST version 1.1 and immune-related RECIST (irRECIST) for solid tumor and the Lugano Classification for non-Hodgkin Lymphoma | 2 Cycles (42 days)
Time to progression (TTP) as assessed by RECIST version 1.1 and immune-related RECIST (irRECIST) for solid tumor and the Lugano Classification for non-Hodgkin Lymphoma | 2 Cycles (42 days)
Disease control rate (DCR) as assessed by RECIST version 1.1 and immune-related RECIST (irRECIST) for solid tumor and the Lugano Classification for non-Hodgkin Lymphoma | 2 Cycles (42 days)
Progression-free survival (PFS) as assessed by RECIST version 1.1 and immune-related RECIST (irRECIST) for solid tumor and the Lugano Classification for non-Hodgkin Lymphoma | 2 Cycles (42 days)
Peak plasma concentration (Cmax) | 2 Cycles (42 days)
Plasma concentration at the end of a dosing interval (Ctrough) | 2 Cycles (42 days)
Time to reach Cmax (Tmax) | 2 Cycles (42 days)
Area under the curve from time zero to the last timepoint (AUC0-last) | 2 Cycles (42 days)
AUC from time zero to infinity (AUC0-∞) | 2 Cycles (42 days)
AUC during a dosing interval (AUCtau) | 2 Cycles (42 days)
Clearance (CL) | 2 Cycles (42 days)
Volume of distribution at steady state (Vss) | 2 Cycles (42 days)
ADA levels for ADG106. | 2 Cycles (42 days)
Serum biomarkers linked to immunomodulation and cytokine release: such as TNFα, IFN-γ, IL 10, IL-6, IL-4, IL-2. | 2 Cycles (42 days)
Cell counts for circulating T, natural killer (NK), and B cells. | 2 Cycles (42 days)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shanghai Dongfang Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma Y, Luo F, Zhang Y, Liu Q, Xue J, Huang Y, Zhao Y, Yang Y, Fang W, Zhou T, Chen G, Cao J, Chen Q, She X, Luo P, Liu G, Zhang L, Zhao H. Preclinical characterization and phase 1 results of ADG106 in patients with advanced solid tumors and non-Hodgkin's lymphoma. Cell Rep Med. 2024 Feb 20;5(2):101414. doi: 10.1016/j.xcrm.2024.101414. Epub 2024 Feb 7. PMID 38330942